CLINICAL TRIAL: NCT03738917
Title: Effectiveness of Antitussives, Anticholinergics and Honey Versus Usual Care in Adults With Uncomplicated Acute Bronchitis.
Brief Title: Effectiveness of Antitussives, Anticholinergics and Honey Versus Usual Care in Adults With Acute Bronchitis.
Acronym: AB4T
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IJG-AB4T-2018
Record Dates: First submitted 2018-11-05; First posted 2018-11-13 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2021-08

CONDITIONS: Acute Bronchitis
Keywords: Cough; Dextromethorphan; Ipratropium; Honey.
MeSH Terms: conditions — Bronchitis; Cough | interventions — Antitussive Agents; Cholinergic Antagonists; Honey; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Multicentre, pragmatic, parallel group, open randomized trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dextromethorphan (Active Comparator): Usual clinical practice + dextromethorphan (15 milligrams unit), one 15 mg-tablet t.i.d. up to a maximum of 14 days.
  Interventions: Drug: Dextromethorphan 15 milligrams
- Ipratropium (Active Comparator): Usual clinical practice + ipratropium bromide 20Micrograms Inhaler each puff), 2 puffs t.i.d. up to a maximum of 14 days.
  Interventions: Drug: Ipratropium Bromide 20Micrograms Inhaler
- Honey (Active Comparator): Usual clinical practice + Honey 30 g (full tablespoon) t.i.d. up to a maximum of 14 days. Patients will be given two 750 milligram bottles of wildflower honey (the most frequent type of honey used in our country) and patients will be recommended to add the honey to a cup of lemon or thyme juice, milk herbal tea, yogurt, as a hot toddy, etc.
  Interventions: Dietary Supplement: Honey 30 g (full tablespoon)
- Usual clinical practice (Placebo Comparator): Usual care.
  Interventions: Other: Usual clinical practice

INTERVENTIONS:
Drug: Dextromethorphan 15 milligrams — This drug is already marketed, and therefore, the manufacturer is responsible for the elaboration and control of samples. This study drug will be provided free to the participants by the sponsor.
  Other Names: Antitussive
  Arms: Dextromethorphan
Drug: Ipratropium Bromide 20Micrograms Inhaler — This drug is already marketed, and therefore, the manufacturer is responsible for the elaboration and control of samples. This study drug will be provided free to the participants by the sponsor.
  Other Names: Anticholinergic
  Arms: Ipratropium
Dietary Supplement: Honey 30 g (full tablespoon) — This study product will be provided free to the participants by the sponsor.
  Other Names: Dietary supplement
  Arms: Honey
Other: Usual clinical practice — Clinicians will not be allowed to prescribe antitussives, including codeine, anticholinergic inhalers and they will not be allowed to recommend the use of honey.
  Other Names: Usual care
  Arms: Usual clinical practice

SUMMARY:
This study, which is aimed at comparing the effectiveness of 3 symptomatic therapies (dextromethorphan, ipratropium and honey) associated with usual care and the usual care in adults with acute bronchitis, is a multicentre, pragmatic, parallel group, open randomised trial. Patients aged 18 or over with uncomplicated acute bronchitis, with cough <3 weeks as the main symptom, scoring ≥ 4 in either daytime or nocturnal cough on a 7-point Likert scale, will be randomised to one of the 4 groups. Sample: 668 patients. The primary outcome will be the number of days with moderate-severe cough.

DETAILED DESCRIPTION:
Despite the frequent use of therapies in acute bronchitis, encouraged by the over-the-counter availability in pharmacies, the evidence of their benefit is scarce, since only a few clinical trials have been published, with low sample sizes, poor methodological quality and mainly in children. The objective of this study is to compare the effectiveness of 3 symptomatic therapies (dextromethorphan, ipratropium and honey) associated with usual care and the usual care in adults with acute bronchitis. This will be a multicentre, pragmatic, parallel group, open randomised trial. Patients aged 18 or over with uncomplicated acute bronchitis, with cough for less than three weeks as the main symptom, scoring ≥ 4 in either daytime or nocturnal cough on a 7-point Likert scale, will be randomised to one of the following four groups: usual care, usual care + dextromethorphan 30 mg t.i.d., usual care + ipratropium bromide inhaler 20 µg 2 puffs t.i.d, or usual care + 30 mg (a spoonful) of honey t.i.d., all taken for up to 14 days. The exclusion criteria will be: pneumonia, criteria for hospital admission, pregnancy or lactation, concomitant pulmonary disease, associated significant comorbidity, allergy, intolerance or contraindication to any of the study drugs, admitted to a long-term residence, or inability to give informed consent. Sample: 668 patients. The primary outcome will be the number of days with moderate-severe cough in the intention-to-treat (ITT) population, i.e., the number of days from the randomisation visit until the last day the patient scores three or more in either daytime or nocturnal cough in the symptom diary. All patients will be given a symptom diary to be self-administered while symptoms are present. A second visit will be scheduled at day 2-3 for assessing evolution, with two more visits at days 15 and 29 for clinical assessment, evaluation of adverse effects, re-attendance and complications. Patients still with symptoms at day 29 will be called six weeks after the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older, and
* symptoms of acute bronchitis with cough starting within 3 weeks before study inclusion, and
* patients who score ≥ 4 in either the daytime and/or nocturnal cough on a 7-point Likert scale, and
* patients who consent to participate.

Exclusion Criteria:

* suspected pneumonia; if the professional suspects pneumonia, a chest X-ray will be recommended and the patient will be randomized if this diagnosis is discarded; or
* criteria for hospital admission (impaired consciousness, respiratory rate > 30 breaths/minute, pulse > 125 beats/minute, systolic blood pressure <90 mm Hg or diastolic blood pressure <60 mm Hg, temperature > 104°F or oxygen saturation <92%)
* pregnancy or breast feeding
* baseline respiratory disease such as chronic obstructive pulmonary disease, asthma, tuberculosis or bronchiectasis
* associated significant comorbidity, such as moderate-severe heart failure, dementia, acute myocardial infarction/recent cerebral vascular accident (< 3 months), severe liver failure, severe renal failure
* immunosuppression, such as chronic infection by HIV, transplanted, neutropenic, or patients receiving immunosuppressive treatment
* active neoplasm
* terminal illness
* history of intolerance or allergy to any of the study treatments
* patients in whom, in the opinion of the investigator, treatment with dextromethorphan, ipratropium bromide or honey is contraindicated
* patients living in long-term institutions
* difficulty in conducting scheduled follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Duration of moderate-severe cough in days in the four arms. | Day 29.
  Number of days until the last day the patient scores 3 in either daytime cough or nocturnal cough in the symptom diary. Each symptom will be scored by the patient on a 7-point Likert scale, which has been used in previous studies (0=not affected; 1=very little problem; 2=slight problem; 3=moderately bad; 4=bad; 5=very bad; 6=as bad as it could be).

SECONDARY OUTCOMES:
Duration of cough in days in the four arms. | Days 15 and 29. If the patient continues to score 2 or more at day 29 will be called at day 43.
  Number of days until the last day the patient scores 2 in either daytime cough or nocturnal cough in the symptom diary. Each symptom will be scored by the patient on a 7-point Likert scale, which has been used in previous studies (0=not affected; 1=very little problem; 2=slight problem; 3=moderately bad; 4=bad; 5=very bad; 6=as bad as it could be).
Duration of moderate-severe daytime cough in days in the four arms. | Days 15 and 29. If the patient continues to score 3 or more at day 29 will be called at day 43.
  Number of days until the last day the patient scores 3 in daytime cough in the symptom diary. This symptom will be scored by the patient on a 7-point Likert scale, which has been used in previous studies (0=not affected; 1=very little problem; 2=slight problem; 3=moderately bad; 4=bad; 5=very bad; 6=as bad as it could be).
Duration of moderate-severe nocturnal cough in days in the four arms. | Days 15 and 29. If the patient continues to score 3 or more at day 29 will be called at day 43.
  Number of days until the last day the patient scores 3 in nocturnal cough in the symptom diary. This symptom will be scored by the patient on a 7-point Likert scale, which has been used in previous studies (0=not affected; 1=very little problem; 2=slight problem; 3=moderately bad; 4=bad; 5=very bad; 6=as bad as it could be).
Duration of moderate-severe symptoms in days in the four arms. | Days 15 and 29. If the patient continues to score 3 or more at day 29 will be called at day 43.
  Number of days until the last day the patient scores 3 in any of the symptoms in the symptom diary. Each symptom will be scored by the patient on a 7-point Likert scale, which has been used in previous studies (0=not affected; 1=very little problem; 2=slight problem; 3=moderately bad; 4=bad; 5=very bad; 6=as bad as it could be).
Duration of severe symptoms in days in the four arms. | Days 15 and 29.
  Number of days until the last day the patient scores 5 in any of the symptoms in the symptom diary. Each symptom will be scored by the patient on a 7-point Likert scale, which has been used in previous studies (0=not affected; 1=very little problem; 2=slight problem; 3=moderately bad; 4=bad; 5=very bad; 6=as bad as it could be).
Duration of symptoms in days in the four arms. | Days 15 and 29. If the patient continues to score 2 or more at day 29 will be called at day 43.
  Number of days until the last day the patient scores 2 in any of the symptoms in the symptom diary. Each symptom will be scored by the patient on a 7-point Likert scale, which has been used in previous studies (0=not affected; 1=very little problem; 2=slight problem; 3=moderately bad; 4=bad; 5=very bad; 6=as bad as it could be).
Duration of moderate-severe cough in days according to the basal degree of bronchial hyper-reactiveness in the four arms. | The peak-flow will be determined at day 1.
  Number of days until the last day the patient scores 3 in either daytime cough or nocturnal cough in the symptom diary. Each symptom will be scored by the patient on a 7-point Likert scale, which has been used in previous studies (0=not affected; 1=very little problem; 2=slight problem; 3=moderately bad; 4=bad; 5=very bad; 6=as bad as it could be). Bronchial hyper-responsiveness will be determined with three peak-flow measurements at day 1 and the highest of three peak flow measurements will be collected.
Percentage of antibiotics and different symptomatic treatments used in the four arms. | Days 2-4, 15 and 29.
  This information will be collected every day by the patients themselves.
Number of days of absence from work in the four arms. | Day 15.
  Electronic records and sick leave certifications.
Patients re-attendance for symptoms related to the episode of acute bronchitis within the first 42 days. | Day 29 and phone call at day 43.
  The number of re-attendances to any doctor regarding the episode of acute bronchitis will be collected from the electronic records.
Number of complications related to the episode of acute bronchitis within the first 28-42 days. | Day 29-43.
  The number of complications will be collected through electronic records and hospital certifications.
Patient satisfaction in the four arms. | Day 15 or 29.
  Patient satisfaction will be collected in the same symptom diaries by the patients themselves by means of questions included in the symptom diary.
Number of adverse events in the four arms. | Days 2-4, 15 and 29.
  The number of adverse events will be collected by the participating doctor by means of questions.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Moragas, MD PhD, Study Chair — Catalan Institute of Health
Locations (12):
- Spain (12):
  - Nova Lloreda Health Center, Badalona, Catalonia
  - Martí i Julià Health Center, Badalona, Catalonia
  - Balaguer Health Center, Balaguer, Catalonia
  - Via Roma Health Centre, Barcelona, Catalonia
  - La Marina Health Center, Barcelona, Catalonia
  - CAP Passeig Maragall (EAP Camp de l'Arpa), Barcelona, Catalonia
  - Cornellà - La Gavarra Health Center, Cornellà de Llobregat, Catalonia
  - Pineda de Mar Health Center, Pineda de Mar, Catalonia
  - Ca n'OriacHealth Center, Sabadell, Catalonia
  - Molí Nou Health Center, Sant Boi de Llobregat, Catalonia
  - Singuerlin Health Center, Santa Coloma de Gramenet, Catalonia
  - CAP Jaume I, Tarragona, Catalonia

IPD SHARING:
Plan to Share IPD: Yes
Reposition of data in Scientia
Supporting Information: Study Protocol, SAP
Time Frame: 2021
Access Criteria: Scientia
URL: http://scientiasalut.gencat.cat

REFERENCES:
- [Derived] Llor C, Moragas A, Ouchi D, Monfa R, Garcia-Sangenis A, Gomez-Lumbreras A, Pera H, Pujol J, Morros R. Effectiveness of antitussives, anticholinergics, and honey versus usual care in adults with uncomplicated acute bronchitis: a multiarm randomized clinical trial. Fam Pract. 2023 Mar 28;40(2):407-413. doi: 10.1093/fampra/cmac112. PMID 36239199
- [Derived] Cots JM, Moragas A, Garcia-Sangenis A, Morros R, Gomez-Lumbreras A, Ouchi D, Monfa R, Pera H, Pujol J, Bayona C, de la Poza-Abad M, Llor C. Effectiveness of antitussives, anticholinergics or honey versus usual care in adults with uncomplicated acute bronchitis: a study protocol of an open randomised clinical trial in primary care. BMJ Open. 2019 May 16;9(5):e028159. doi: 10.1136/bmjopen-2018-028159. PMID 31101700